CLINICAL TRIAL: NCT03733197
Title: Developing a Barbershop-Based Trial on Masculinity Barriers to Care and Colorectal Cancer Screening Uptake Among African-American Men Using a Mixed Methods Approach
Brief Title: #CuttingCRC: Barbershop-Based Trial & Colorectal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer employed at institutuion
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Dr. Charles R. Rogers, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00113679
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Mixed Methods Approach
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culture specific (Experimental): The culture-specific arm "may" entail FIT kits plus barbers as motivational interviewers.
  Interventions: Behavioral: Culture Specific
- Control (Experimental): Distribution of CRC screening brochures & FIT (Fecal Immunochemical Test) kits by barbers
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Culture Specific — We anticipate the culture-specific arm developed minimally will include two core components: barbers as motivational interviewers, and (2) fecal immunochemical test (FIT) kits distributed by barbers. If we choose this route for the culture-specific arm, preliminary data from our barbers suggest I teach the barbers the MI technique using content that stems from Aim 1 findings. Additional components for this arm may be developed during the APEASE process.
  Arms: Culture specific
Behavioral: Control — the (control) arm will include an informational CRC screening brochure developed by the American Cancer Society plus a FIT kit distributed by the barbers.
  Arms: Control

SUMMARY:
The goal of this behavior change focused, culture-specific, pilot, peer intervention is to target masculinity barriers to medical care (MBMC) considering a range of psychosocial factors associated with uptake of CRC screening (fecal immunochemical test (FIT)) among African-American men. Barbershops will serve as intervention sites and barbers will be trained in the technique of Motivational Interviewing (MI) which will guide the barbers to encourage their clients with culturally relevant messaging to take a FIT kit home and then send to the lab for processing (uptake). The main questions it aims to answer are the feasibility of recruitment, sample size estimation, preliminary efficacy, and the acceptability of barbers to deliver culture-specific messages that aim to overcome masculinity barriers to medical care.

Researchers will compare the culture-specific intervention with a control arm, where barbers provide their client an evidenced-based American Cancer Society brochure on colorectal cancer screening to understand if barbers peers using MI and culturally relevant messaging better overcome masculinity barriers to medical care than the barber using the brochure alone.

DETAILED DESCRIPTION:
The purpose of Dr. Rogers' research plan involves developing and pilot testing a theory-driven, culture-specific intervention that specifically targets masculinity barriers to medical care and colorectal cancer (CRC) uptake among African-American men (ages 45-75). CRC is preventable as screening leads to identification and removal pre-cancerous polyps; however, African-American men consistently have the highest CRC mortality rates across all gender and racial/ethnic groups; and their CRC screening uptake remains low for uncertain reason. Contributing factors are etiologically complex, yet but culture-specific masculinity barriers to care may contribute to low CRC screening uptake among African-American men. Examining masculinity barriers to care is vital as CRC screening may challenge some cultural role expectations and self-representations of African-American men whose tendency is to delay help-seeking medical care. The study's specific aims are to: 1) develop, validate, and test a culture specific measure of masculinity barriers to medical care relative to CRC screening uptake among African-American men; and 2) develop and pilot test a theory-driven, culture-specific intervention that targets masculinity barriers to medical care, psychosocial factors, and CRC screening uptake among African-American men. Barbershops are historically known as culturally appropriate and trusted venues in African-American communities, and are critical for this research as they provide a pathway for reaching African-American men with masculinity barriers to care who are not regularly receiving healthcare services, and in particular, CRC screening. This study and integrated training plan well-position Dr. Rogers to launch an independent investigator career focused on informing culture-specific interventions to eliminate cancer inequities among African-American men.

The investigator will conduct research in the metro areas of Salt Lake City (Salt Lake City-Provo-Orem) of Utah; Minneapolis-St. Paul, Minnesota; Columbus, Ohio; and Milwaukee, Wisconsin. African American men's CRC screening rates in UT and Wisconsin are substantially lower than in other states, and the aforementioned metro regions have the largest population of African-Americans in each state. Approach. The investigator proposes a multi-stage mixed methods study (Figure 1), beginning with an exploratory sequential design validating the items for subsequent use in a pilot mixed methods intervention to accomplish aims. For Aim 1 (Years 1-2), the investigator collected and analyzed QUALitative data from 2 sources - focus groups and cognitive interviews - to validate and test a culture-specific scale of masculinity barriers to medical care among African-American men (hereafter called the Masculinity Barriers to Care Scale, MBCS). Next, the investigator administered the MBCS as an online QUANTtitative survey with the target population to evaluate the association between scale scores and CRC screening uptake. For Aim 2 (Years 3-6), the investigator will consider existing evidence-based approaches (e.g., motivation interviewing), the integrated results (QUAL + QUANT) from Aim 1 regarding masculinity barriers to care, and community input to design a novel, culture specific, behavioral intervention - one aimed at increasing CRC screening uptake (fecal immunochemical test; FIT) among African-American men and feasible for delivery in barber shops. The investigator will pilot test the peer intervention in a two-arm cluster randomized intervention (6 barbershops, randomized by site-2 shops in each state, specifically, Wisconsin, Ohio, and Minnesota) to account for differences in barbershop culture and reduce contamination. The primary outcomes for the pilot are recruitment, sample size estimation, preliminary efficacy, and acceptability. The investigator will also conduct post-intervention interviews with participants from both arms to evaluate acceptability (i.e., why and how each arm was or was not successful).

ELIGIBILITY:
Characteristics of Participants/Inclusion Criteria:

[Phase 1 of 2]

* Aim 1A: men who 1) self-identified as non-Hispanic Black/African American, 2) were born in the US; 3) were between ages 45-75; 4) had a working telephone; 5) spoke and understood English; & 6) resided in Utah, Ohio, or Minnesota.
* Aim 1B: men who 1) self-identified as non-Hispanic Black/African American, 2) were born in the US; 3) were between ages 45-75; 4) had a working telephone; 5) spoke and understood English; 6) resided in Utah, Ohio, or Minnesota; & 7) had a phone with internet capabilities.

Participant Exclusion Criteria:

[Phase 1 of 2]

* Aim 1A: men who 1) did not self-identify as non-Hispanic Black/African American, 2) were not born in the US; 3) were not between ages 45-75; 4) did not have a working telephone; 5) did not speak and understand English; & 6) did not reside in Utah, Ohio, or Minnesota.
* Aim 1B: men who 1) did not self-identify as non-Hispanic Black/African American, 2) were not born in the US; 3) were not between ages 45-75; 4) did not have a working telephone; 5) did not speak or understand English; 6) did not reside in Utah, Ohio, or Minnesota; & 7) did not have a phone with internet capabilities.

[Phase 2]

Inclusion: For Aim 2, our pilot intervention Eligibility Criteria & Recruitment includes 60 non-Hispanic Black/African-American male participants who: 1) have never completed CRC screening; 2) are 45-75 years old; 3) were born in the U.S.; 4) reside in Minnesota, Ohio, or Wisconsin; 5) have a telephone with internet, and 6) speak English. As a feasibility intervention, sample size is not based on the power to detect a certain effect size. Rather, n = 60 (30 per arm) was chosen based on practical considerations (e.g., cost, recruitment). With the assistance of barbers and culture-specific marketing materials, we will recruit at least five participants per week from six intervention participation sites (barbershops).

[Phase 2]

Exclusion: For Aim 2, our pilot intervention Eligibility Criteria & Recruitment excludes men who are not Non-Hispanic Black/African-American as well as those who: 1) have never completed CRC screening; 2) are not 45-75 years old; 3) were not born in the U.S.; 4) do not reside in Minnesota, Ohio, or Wisconsin; 5) do not have a telephone with internet, and 6) do not speak English.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self described as male
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Scale development | Year 1-2
  Develop, validate, and test a culture-specific measure of masculinity barriers to medical care relative to psychosocial factors and CRC screening uptake among African-American men

SECONDARY OUTCOMES:
Pilot intervention | Year 3-6
  Develop and pilot test a theory-driven, culture-specific intervention that targets masculinity barriers to medical care, psychosocial factors, and CRC screening update among African-American men.

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Rogers, PhD, MPH, MS, Principal Investigator — Medical College of Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Sharing de-identified participant data stemming from focus groups, cognitive interviews, surveys, intervention arms, and post trial interviews.
Time Frame: Years 1-5
URL: https://cuttingcrc.com

REFERENCES:
- [Derived] Rogers CR, Okuyemi K, Paskett ED, Thorpe RJ Jr, Rogers TN, Hung M, Zickmund S, Riley C, Fetters MD. Study protocol for developing #CuttingCRC: a barbershop-based trial on masculinity barriers to care and colorectal cancer screening uptake among African-American men using an exploratory sequential mixed-methods design. BMJ Open. 2019 Jul 24;9(7):e030000. doi: 10.1136/bmjopen-2019-030000. PMID 31345981